CLINICAL TRIAL: NCT00759148
Title: Moxifloxacin AF Ophthalmic Solution for Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-40
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Bacterial Conjunctivitis
Keywords: pink eye; conjunctivitis; moxifloxacin; fluoroquinolone
MeSH Terms: conditions — Conjunctivitis, Bacterial; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin AF (Experimental): Moxifloxacin Alternative Formulation (AF) Ophthalmic Solution 0.5%, 1 drop in each eye twice daily for 3 days
  Interventions: Drug: Moxifloxacin Alternative Formulation (AF) Ophthalmic Solution 0.5%
- Vehicle (Placebo Comparator): Moxifloxacin AF vehicle, 1 drop in each eye twice daily for 3 days
  Interventions: Other: Moxifloxacin AF Vehicle

INTERVENTIONS:
Drug: Moxifloxacin Alternative Formulation (AF) Ophthalmic Solution 0.5% — Eye drops
  Arms: Moxifloxacin AF
Other: Moxifloxacin AF Vehicle — Inactive ingredients used as a placebo for masking purposes
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Moxifloxacin AF Ophthalmic Solution compared to Moxifloxacin AF Vehicle in the treatment of bacterial conjunctivitis in patients one month of age or older.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bacterial conjunctivitis in 1 or both eyes;
* Able to understand and sign an informed consent form. If subject is <18 years of age, the informed consent must be understood and signed by the subject's legally authorized representative;
* Agrees to comply with the visit schedule and other requirements of the study;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Signs and symptoms of bacterial conjunctivitis for longer than 4 days prior to Day 1;
* Presence of concomitant viral infection;
* Infants with ophthalmia neonatorum of gonococcal, Chlamydia, herpetic or chemical origin;
* Infants whose birth mothers had any sexually transmitted disease within 1 month prior to delivery;
* Infants undergoing treatment for retinopathy of prematurity;
* Contact lens wear during the course of the study;
* Only 1 sighted eye or vision in either eye not correctable to 0.6 logMAR units (20/80) or better;
* Use of medications, as specified in the protocol;
* Any systemic or ocular disease or disorder, complicating factors or structural abnormality that could negatively affect the conduct or outcome of the study;
* Known or suspected allergy or hypersensitivity to fluoroquinolones;
* Pregnant, lactating, or of childbearing potential and not using adequate birth control to prevent pregnancy;
* Other protocol-specified exclusion criteria may apply.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Ltd., Study Director — Alcon Research

REFERENCES:
- [Derived] Tauber S, Cupp G, Garber R, Bartell J, Vohra F, Stroman D. Microbiological efficacy of a new ophthalmic formulation of moxifloxacin dosed twice-daily for bacterial conjunctivitis. Adv Ther. 2011 Jul;28(7):566-74. doi: 10.1007/s12325-011-0037-x. Epub 2011 Jun 14. PMID 21681652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 108 study centers located in the US.
Pre-assignment Details: 1179 subjects with bacterial conjunctivitis were randomized and treated to Moxifloxacin AF or Moxifloxacin AF vehicle.
Period: Overall Study
Arm/Group | Moxifloxacin AF | Vehicle
Started | 593 | 586
Completed | 579 | 554
Not Completed | 14 | 32
Not completed — Adverse Event | 1 | 6
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Lost to Follow-up | 3 | 9
Not completed — Treatment Failure | 6 | 10
Not completed — Reason not given | 1 | 0

BASELINE CHARACTERISTICS:
Population: This population analysis includes all subjects who received study drug (Safety Analysis Set).
Groups:
- Moxifloxacin AF: Moxifloxacin AF Ophthalmic Solution 0.5%, 1 drop in each eye twice daily for 3 days
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin AF | Vehicle | Total
Number analyzed (Participants) | 593 | 586 | 1179
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 49 | 47 | 96
  Children (2-11 years) | 174 | 184 | 358
  Adolescents (12-17 years) | 71 | 72 | 143
  Adults (18-64 years) | 257 | 230 | 487
  From 65-84 years | 38 | 48 | 86
  85 years and over | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 353 | 338 | 691
  Male | 240 | 248 | 488

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure at the Day 4 (EOT)/Exit Visit
Description: Clinical cure was attained if the sum of the 2 cardinal ocular signs of bacterial conjunctivitis (bulbar conjunctival injection and conjunctival discharge/exudate) was zero (ie, normal or absent) 12-48 hours after the last dose. Clinical cure was reported as a percentage. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 4
Population: This analysis population includes all patients who received drug, had at least 1 on-therapy visit and were pathogen positive for bacteria on Day 1 (Microbiological Intent-to-Treat (MBITT) Analysis Set).
Measure: Number; unit: percentage of subjects
Arm/Group | Moxifloxacin AF | Vehicle
Number analyzed (Participants) | 424 | 423
percentage of subjects | 62.5 | 50.6

2. Secondary Outcome: Microbiological Success at the Day 4 (EOT)/Exit Visit
Description: Microbiological success was attained if the pre-therapy bacterial pathogens were eradicated 12-48 hours after the last dose. Microbiological success is reported as a percentage. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 4
Population: MBITT Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Moxifloxacin AF | Vehicle
Number analyzed (Participants) | 424 | 423
percentage of subjects | 74.5 | 56

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 4 days
Description: An AE was defined as any untoward change (expected or unexpected) in a patient's ophthalmic and/or medical health that occurred after initiation of study treatment. AEs were obtained as solicited comments from the study patient/guardian and as observations by the study investigator.
Groups:
- Moxifloxacin AF: Subjects exposed to Moxifloxacin AF
- Vehicle: Subjects exposed to Moxifloxacin AF Vehicle
Arm/Group | Moxifloxacin AF | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/593 | 0/586
Serious Adverse Events (participants affected / at risk) | 0/593 | 0/586
Other Adverse Events (participants affected / at risk) | 0/593 | 0/586

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review study related information prior to presentation or publication.